CLINICAL TRIAL: NCT02128269
Title: An Open-Label Proof of Concept Phase IIa Trial of ALXN1007 for the Treatment of Non-criteria Manifestations of Antiphospholipid Syndrome
Brief Title: Phase IIa Trial of ALXN1007 for the Treatment of Non-criteria Manifestations of Antiphospholipid Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Screening discontinued early due to slow patient enrollment
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1007-APS-201; 2013-003588-73 (EudraCT Number)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: Antiphospholipid (aPL)-Positive
Keywords: Antiphospholipid (aPL)-positive; Antiphospholid syndrome (APS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ALXN1007- Open label study (Experimental): ALXN1007
  Interventions: Biological: Study Drug- ALXN1007

INTERVENTIONS:
Biological: Study Drug- ALXN1007 — 10 mg/kg IV q 2 weeks x 12 doses

SUMMARY:
The primary purpose of this study was to evaluate the safety and tolerability of intravenous (IV) ALXN1007 in persistently antiphospholipid (aPL)-positive patients with at least 1 of the following non-criteria manifestations of APS: aPL-nephropathy, skin ulcers and/or thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

Patients with a persistent and clinically significant aPL profile

Patients with at least 1 of the following non-criteria manifestations of APS:

1. aPL-nephropathy (diagnosed by kidney biopsy within 12 months of Screening) confirmed based on the updated APS Classification Criteria recommendations, and urine protein to creatinine ratio > 1.0 at the time of the Screening visit and/or
2. Skin ulcers (non-infected livedoid vasculitis-like skin ulcer and/or large skin ulceration resembling pyoderma gangrenosum) for at least 4 weeks prior to the Screening visit, diagnosed by physical examination, and/or
3. Persistent active thrombocytopenia (diagnosed by platelet counts <100 x 103/μL and ≥20 x 103/μL [SI: <100 x 109/L and ≥ 20 x 109/L]) and confirmed at the time of screening (at least 4 weeks after previous test) based on the updated APS Classification Criteria recommendations Patients and spouse/partner who is of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (at least 1 of which must be a barrier method) starting at Screening and continuing through the entire study.

Patients with aPL-nephropathy must be receiving or agree to initiate an ACE inhibitor or angiotensin receptor blocker at least 4 weeks prior to initiation of ALXN1007 treatment; unless patient is documented to be intolerant. Patients receiving oral corticosteroids must be on a stable dose of ≤ 10 mg/day of prednisone or equivalent dose of another corticosteroid preparation for at least 4 weeks prior to the first dose of ALXN1007. Patients receiving immunosuppressive medications (including but not limited to methotrexate, hydroxychloroquine, azathioprine, cyclosporine and mycophenolate mofetil) must be on a stable dose for at least 4 weeks prior to the first dose of ALXN1007. Patients receiving oral anticoagulants or antiplatelet agents (including but not limited to aspirin) must be on stable doses for at least 4 weeks prior to first dose of ALXN1007.

Patients must be willing and able to give written informed consent and to comply with all study visits and procedures.

Exclusion Criteria:

Patients meeting the ACR classification criteria for systemic lupus erythematosus, systemic sclerosis or other systemic autoimmune diseases other than Primary APS.

Patients experiencing an acute thrombosis or a Major Adverse Vascular Event (MAVE) within 12 weeks prior to first administration of ALXN1007.

Patients with skin ulcers from causes other than aPL or who are positive for DVT or venous insufficiency at Screening. Patients with renal function status requiring chronic dialysis (defined as dialysis on a regular basis as renal replacement therapy). Patients with unresolved meningococcal disease or with known active bacterial, viral, fungal, mycobacterial or other infection. Patients that have received IVIg treatment within 4 weeks prior to first dose of ALXN1007. Patients that have received a course of rituximab (RITUXAN®) therapy within 12 months prior to first dose of ALXN1007 or have evidence of persistent depletion of the targeted lymphocyte population. Women who are pregnant or nursing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bert Yao, M.D., Ph.D., Study Director — Alexion Medical Monitor
Locations (9):
- United States (3):
  - Hospital for Special Surgery, New York, New York
  - University of Texas Medical Branch, Galveston, Texas
  - O & O Alpan, LLC, Fairfax, Virginia
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil
- France (2):
  - Hôpital Cochin, Paris, France 75679
  - Hopital Claude Huriez - CHU Lille, Lille, Nord
- Azienda Ospedaliera di Padova, Padua, Italy
- Hokkaido University Hospital, Sapporo, Hokkaido 060-8648, Japan
- University College London Hospitals, London, Greater London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- ALXN1007: ALXN1007 10 mg/kg IV q 2 weeks x 12 doses
Period: Treatment Period
Arm/Group | ALXN1007
Started | 9
Completed | 7
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Period: Follow-up
Arm/Group | ALXN1007
Started | 9 (All enrolled patients were followed for 12 weeks after their last infusion of ALXN1007.)
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ALXN1007- Open Label Study: ALXN1007
  ALXN1007: 10 mg/kg IV q 2 weeks x 12 doses
Arm/Group | ALXN1007- Open Label Study
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4
  Japan | 2
  Italy | 1
  France | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Intravenous (IV) ALXN1007 as Measured by Percentage of Patients Reporting Adverse Events
Time Frame: Treatment Period (24 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | ALXN1007
Number analyzed (Participants) | 9
Participants | 8

ADVERSE EVENTS:
Time Frame: Treatment Period (24 weeks) and Follow-up Period (12 weeks).
Arm/Group | ALXN1007- Open Label Study
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN1007- Open Label Study (N=9)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Cholestasis (Hepatobiliary disorders) | 1
Liver Cytolysis (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALXN1007- Open Label Study (N=9)
Anaemia (Blood and lymphatic system disorders) | 1
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Bronchitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral Herpes (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Staphylococcal Infection (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 4
Urethritis (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Varicose vein (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication rights are tied to the completion of the multi-center publication